CLINICAL TRIAL: NCT02137967
Title: Clinical Evaluation of Sodium Hypochlorite Pulpotomies in Primary Molars: A Long-Term Follow-Up in Comparison With Conventional 20% Formocresol Pulpotomies
Brief Title: Sodium Hypochlorite Pulpotomies in Primary Molars: Comparison With Conventional 20% Formocresol Pulpotomies
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201105091RB
Record Dates: First submitted 2012-01-02; First posted 2014-05-14 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Dental Pulp Disease
MeSH Terms: conditions — Dental Pulp Diseases | interventions — formocresol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- NaOCl pulpotomy (Experimental): Use 2.5% NaOCl as pulpotomy medication
  Interventions: Procedure: NaOCl pulpotomy; Drug: 2.5% NaOCl
- FC pulpotomy (Active Comparator): Use 20% Formocresol as pulpotomy medicament
  Interventions: Procedure: FC pulpotomy; Drug: 20% Formocresol

INTERVENTIONS:
Procedure: NaOCl pulpotomy — Use 2.5% NaOCl as pulpotomy medicament for primary molars
  Arms: NaOCl pulpotomy
Procedure: FC pulpotomy — Use 20% Formocresol as pulpotomy medicament for primary molars
  Arms: FC pulpotomy
Drug: 2.5% NaOCl
  Arms: NaOCl pulpotomy
Drug: 20% Formocresol
  Arms: FC pulpotomy

SUMMARY:
Formocresol (FC) is the most universally taught and most widely used pulpotomy medicament in the primary teeth. However, concerns have been raised over the use of FC because of its toxicity and potential carcinogenicity. A substitution for FC has been investigated but evidence is lacking to conclude which is the most appropriate technique for pulpotomies in primary teeth. Sodium hypochlorite (NaOCl) has been used in root canal irrigant for more than 80 years, and it is at present the most popular irrigant in root canal treatment. Studies have showed that NaOCl is biological compatible and is a very good antimicrobial solution without being a pulpal irritant. Recent studies using sodium hypochlorite as pulpotomy medicament in primary molars showed promising results. In this project, the investigators propose a randomized clinical trial, which will be performed in Pediatric Dentistry Department of the National Taiwan University Hospital, to compare the treatment outcomes between NaOCl and FC in human primary molars needing pulpotomy treatment. The aim of this sudy is to determining weather NaOCl is a suitable replacement for FC in the pulpotomy of human primary molar teeth. To assess this aim, 200 healthy children from 2.5 to 9 year-old, who have at least one primary first or second molars diagnosed to receive pulpotomy treatment will be recruited in this project. The involved teeth will be randomly assigned to the control group (dilute 20% Formocresol (DFC)) or experimental group (2.5% NaOCl). At 3, 6, 9, 12, 15, 18, 21 and 24 months post-treatment, the randomly assigned teeth will be clinically and radiographically evaluated by blinded independent evaluators to the treatment group. The differences will be statistically analyzed using chi-square test, Fisher exact test, and t-test, using a statistical significance at p<0.05.

DETAILED DESCRIPTION:
As Brief summary.

ELIGIBILITY:
Inclusion Criteria:

* healthy, American Society of Anesthesiologists (ASA) Physical Status classification system class I children
* age between 2.5 and 9 years old
* with one or more primary molars need pulpotomy treatment

Exclusion Criteria:

* children younger than 2.5 or older than 9 years of age

Ages: 30 Months to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-09 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change of Clinical Findings | At 3, 6, 9, 12, 15, 18, 21 and 24 months post-treatment
  The outcome will be assessed first by clinical findings. We can discriminate the result are successful or not by scoring the clinical finding from 1 to 4 .
  Criteria for clinical scoring
  1. Asymptomatic, clinical score=1
  2. Slight discomfort: percussion sensitivity; mobility>1mm but<2mm, clinical score=2
  3. Minor discomfort :long-lasting chewing sensitivity; gingival swelling; periodontal pocket formation without exudate; mobility>2mm but<3mm, clinical score=3
  4. major discomfort: Late pathological changes; spontaneous pain; periodontal pocket formation with exudate; sinus tract; mobility≧3 mm; premature tooth loss due to pathology, clinical score=4

SECONDARY OUTCOMES:
Change of Radiographic Findings | At 3, 6, 9, 12, 15, 18, 21 and 24 months post-treatment
  The outcome will be assessed then by radiographic findings. We can discriminate the result are successful or not by scoring the radiographic findings from1 to 5.
  Criteria for radiographic scoring
  1. Dentinal bridge, clinical score=1, regeneration tissue response
  2. No change, clinical score=2, no pathological changes
  3. Pulp canal obliteration, clinical score=3, slight pathological changes, no clinical significance
  4. Periodontal ligament widening, clinical score=3, slight pathological changes, no clinical significance
  5. Internal root resorption (non-perforated), clinical score=4, minor pathological changes
  6. External root resorption, clinical score=4, minor pathological changes
  7. Internal root resorption (perforated), clinical score=4, minor pathological changes
  8. Peri-radicular lesion, clinical score=5, major pathological changes, treatment needed

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Hua Chang, phD, Principal Investigator — Assistant Professor
Locations (1):
- Pediatric dental department, National Taiwan University Hospital, Taipei, Taiwan